CLINICAL TRIAL: NCT06061146
Title: Tislelizumab Combined With Concurrent Chemoradiation Versus Concurrent Chemoradiation for Older Patients With Inoperable Locally Advanced Esophageal Squamous Cell Carcinoma: a Randomized, Parallel-controlled, Multicenter Phase II Clinical Study
Brief Title: Tislelizumab Plus Concurrent Chemoradiation in Older With ESCC
Acronym: TCRTOE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Shanxi Province Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Hunan Cancer Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230954
Record Dates: First submitted 2023-09-10; First posted 2023-09-29 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: Old Age; Esophageal Cancer; Tislelizumab; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; S 1 (combination); Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Tislelizumab + S1 + Radiotherapy Drug: Tirellizumab IV infusion，200 mg/3w, for 1 year
  Drug: S1 PO, 40~60mg，BID（d1-14，d22-35，two cycles）
  Radiation: Radiation Concurrent Radiation, 1.8Gy/f, 28f
  Interventions: Drug: Arm A; Radiation: Arm A
- Arm B (Active Comparator): S1 + Radiotherapy
  Drug: S1 PO, 40~60mg，BID（d1-14，d22-35，two cycles）
  Radiation: Radiation Concurrent Radiation, 1.8Gy/f, 28f
  Interventions: Drug: Arm B; Radiation: Arm B

INTERVENTIONS:
Drug: Arm A — anti-PD-1 immunotherapy
  Other Names: Tislelizumab
  Arms: Arm A
Drug: Arm A — chemotherapy
  Other Names: S1
  Arms: Arm A
Radiation: Arm A — Radiation Concurrent Radiation, 1.8Gy/f, 28f
  Other Names: Radiotherapy
  Arms: Arm A
Drug: Arm B — chemotherapy
  Other Names: S1
  Arms: Arm B
Radiation: Arm B — Radiation Concurrent Radiation, 1.8Gy/f, 28f
  Other Names: Radiotherapy
  Arms: Arm B

SUMMARY:
This study was conducted in elderly (≥70 years old) patients with locally advanced esophageal squamous cell carcinoma. Aim to find the difference in efficacy and safety between tirilizumab combined with concurrent chemoradiation and standard concurrent chemoradiation.

Concurrent chemoradiation is the standard treatment for elderly esophageal cancer. Tirelizumab is the first-line and second-line standard treatment for advanced esophageal squamous carcinoma. However, the effect of tirilizumab combined with concurrent chemoradiation for elder with locally advanced esophageal squamous cell carcinoma is unkown.

In the study, the investigators plan to enroll 136 elderly subjects with locally advanced esophageal cancer from five hospitals in China. The enrolled patients will be randomly divided into two groups: tirilizumab combined with concurrent chemoradiation group (Tislelizumab + radiotherapy + tigio) and concurrent chemoradiation group (radiotherapy + tigio). The treatment efficiency and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate, cooperated with follow-up visits;
2. Aged ≥ 70 years, both male and female;
3. Histologically confirmed cT1N2-3M0 or cT2-4bN0-3M0 or cT1-4bN0-3M1(supraclavicular lymph node metastasis) locally advanced ESCC (8th AJCC );
4. Clinically staged as II-IVb inoperable locally advanced ESCC(including non-resectable, or with contraindications to or refusal of surgery);
5. ECOG performance status 0 or 1;
6. Presence of measurable and/or non-measurable lesions as defined by RECIST 1.1;
7. Haven't received any previous systemic anti-tumor therapy (including but not limited to systemic chemotherapy, radiotherapy, molecularly targeted drug therapy, immunotherapy, biologic therapy, topical therapy and other investigational therapeutic agents);
8. Provide fresh or archived tumour tissue samples within 6 months (fresh samples preferred) for biomarker analysis (e.g.PD-L1). Sample types are formalin-fixed, paraffin-embedded [FFPE] tumour tissue blocks or at least 5 unstained, 3-5 μm thick FFPE tumour tissue sections;
9. Expected survival ≥ 3 months;
10. Adequate hematologic function, defined as ANC ≥1500/μl, platelet count ≥100,000/μl and hemoglobin count ≥9.0 g/dl or ≥5.6 mmol/l;
11. Adequate renal function, defined as creatinine ≤1.5× ULN or measured or calculated creatinine clearance ≥60 mL/min for those with creatinine levels >1.5× ULN (Calculated from the Cockcroft-Gault formula);
12. Adequate hepatic function, defined as total bilirubin ≤1.5× ULN and ALT/AST/AKP levels ≤2.5× ULN and albumin ≥2.8 g/dl;
13. Adequate coagulation function, defined as INR ≤1.5× ULN and APTT≤1.5× ULN unless the patient is receiving anticoagulant therapy as long as INR is within the therapeutic range;
14. Documented informed consent.

Exclusion Criteria:

1. Surgery for esophageal cancer;
2. Esophageal fistulae due to infiltration of the primary tumour;
3. Risk of gastrointestinal bleeding, oesophageal fistula or oesophageal perforation
4. Poor nutritional status, weight loss of ≥10% in the previous 2 months, with no significant improvement after nutritional intervention;
5. Major surgery or severe trauma within 4 weeks prior to first use of study drug;
6. Uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
7. Received or receiving any of the following treatments in the past:

   1. Anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy or targeted therapy;
   2. Participation in a study of an investigational agent or device within 4 weeks before the first dose of study treatment;
   3. Systemic treatment with corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressive agents is required for 2 weeks before the first dose of study treatment(except for the use of corticosteroids for local inflammation of the oesophagus and for the prevention of allergy and nausea and vomiting). Other special circumstances need to be communicated to the sponsor.Inhaled or topical steroids and adrenocorticotropic hormone replacement at doses >10mg/day prednisone efficacy dose are permitted if the patient does not have active autoimmune disease;
   4. Received an anti-tumour vaccine or received a live vaccine within 4 weeks before the first dose of study treatment;
8. Any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism);Except for patients with vitiligo or those who had asthma or allergies in childhood but did not need any intervention as adults; patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes mellitus treated with stable doses of insulin may be included;
9. Diagnosis of immunodeficiency, including positive HIV test,other acquired/congenital immunodeficiency diseases, organ transplantation and allogeneic bone marrow transplantation;
10. Diagnosis of uncontrolled cardiac clinical symptoms or disease such as a.NYHA II or above heart failure b.unstable angina c.myocardial infarction within 1 year d.clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
11. Severe infections (CTC AE > Grade 2), such as severe pneumonia requiring hospitalisation, bacteraemia, infectious co-morbidities, etc., within 4 weeks before the first use of study treatment; Baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks before the first use of study treatment, except for prophylactic antibiotic use;
12. History of interstitial lung disease or non-infectious pneumonia, or pulmonary insufficiency ≥ grade 3 as confirmed by pulmonary function tests;
13. Active tuberculosis infection detected by history or CT examination, or history of active tuberculosis infection within 1 year before enrollment or more than 1 year previously without regular treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection);
15. Presence of abnormal sodium, potassium, and calcium laboratory test values greater than Grade 1 within 2 weeks prior to randomisation that do not improve with treatment;
16. Known hypersensitivity to large protein preparations, or to any of the components of tirilizumab, or anaphylaxis, hypersensitivity, or contraindication to paclitaxel or cisplatin or to any of the components used within their preparations;

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to 2 years
  overall survival
ORR | up to 2 years
  overall response rate
DoR | up to 2 years
  Duration of Response
AE | up to 3 years
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Zhang, M.D, Principal Investigator — Tian jin cancer hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang K, Wang Q, Cao J, Fan C, Shen W, Xiao Q, Ge X, Zhang T, Liu X, Chen X, Dong J, Li Z, Zheng Z, Yan C, Wang P, Pang Q, Zhang W. Tislelizumab plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy for elderly patients with inoperable locally advanced esophageal squamous cell carcinoma: a multicenter, randomized, parallel-controlled, phase II clinical trial. BMC Cancer. 2025 Feb 25;25(1):347. doi: 10.1186/s12885-025-13758-0. PMID 40001034